CLINICAL TRIAL: NCT00002981
Title: 11C-Methionine and 2-18F-Fluoro-2-Deoxy-D-Glucose PET Imaging in Patients With Progressive Prostate Cancer
Brief Title: PET Scan in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 97-007; P30CA008748 (NIH); MSKCC-97007; NCI-G97-1232
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; carbon-11 methionine

ARMS (1):
- PET Scan (Experimental): Each patient receives C11-methionine intravenously. PET imaging begins immediately after injection for approximately 60 minutes total using standard imaging procedures. Immediately following the completion of imaging after C11-methionine administration, each patient receives FDG intravenously. PET imaging begins approximately 45 minutes thereafter for approximately 60 minutes using standard imaging procedures.
  Interventions: Procedure: positron emission tomography; Radiation: fludeoxyglucose F 18; Radiation: methionine C 11

INTERVENTIONS:
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18
Radiation: methionine C 11

SUMMARY:
RATIONALE: New imaging procedures, such as PET scan, may improve the ability to detect new or recurrent prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Measure the pharmacokinetics, whole body retention of isotope, and biodistribution of C11-methionine and FDG by PET imaging and serial sampling of blood in men with progressive prostate cancer.
* Explore metabolism of each PET scan by comparing the sensitivity of C11-methionine or FDG by PET scanning in androgen independent prostate cancer metastases with the sensitivity of C11-methionine or FDG in androgen dependent metastases on a site by site basis.
* Compare C11-methionine and FDG PET scanning to standard of care diagnostic studies which include the Tc 99m bone scan, computed tomography, and magnetic resonance imaging.

Patients fast for 6 hours prior to PET imaging with the exception of liberal water intake which is encouraged. A two way catheter is placed in the urinary bladder, and continuous isotonic saline irrigation is performed throughout scan acquisition to reduce the interference in imaging lesions in the pelvic lymph nodes and adjacent pelvic bones caused by radiation excreted in urine held in the bladder.

Each patient receives C11-methionine intravenously. PET imaging begins immediately after injection for approximately 60 minutes total using standard imaging procedures. Immediately following the completion of imaging after C11-methionine administration, each patient receives FDG intravenously. PET imaging begins approximately 45 minutes thereafter for approximately 60 minutes using standard imaging procedures.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate adenocarcinoma
* Must have an at least 50% increase in PSA which is sustained for a minimum of 3 observations obtained at least 1 week apart
* Must have development of new lesions on bone scintigraphy or greater than 50% increase in measurable disease on CT or MRI scan
* Metastatic disease

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky greater than 60%

Hematopoietic:

* ANC greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No clinically significant cardiac disease

Pulmonary:

* No clinically significant pulmonary disease

Other:

* No active infection not controlled by antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 0 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 1997-01; Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Larson, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- PET Scan: Each patient receives C11-methionine intravenously. PET imaging begins immediately after injection for approximately 60 minutes total using standard imaging procedures. Immediately following the completion of imaging after C11-methionine administration, each patient receives FDG intravenously. PET imaging begins approximately 45 minutes thereafter for approximately 60 minutes using standard imaging procedures.
  positron emission tomography
  fludeoxyglucose F 18
  methionine C 11
Period: Overall Study
Arm/Group | PET Scan
Started | 173
Completed | 167
Not Completed | 6
Not completed — Inevaluable | 6

BASELINE CHARACTERISTICS:
Arm/Group | PET Scan
Number analyzed (Participants) | 173
Age, Continuous [Median (Full Range); unit: years] | 68 [46 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 160
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 173

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: Up to 9 years
Measure: Median (Full Range); unit: weeks
Arm/Group | PET Scan
Number analyzed (Participants) | 173
weeks | 91.6 [56 to 433]

2. Primary Outcome: Metabolism
Time Frame: 3 years
Population: N/A data were not collected
Arm/Group | PET Scan
Number analyzed (Participants) | 0

3. Primary Outcome: Percentage of Unbiopsied Lesions That Are Confirmed Positive
Description: Comparison of the sensitivity of PET imaging with FDG with standard of care diagnostic methods
Time Frame: 3 years
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Unbiopsied Lesions
Arm/Group | PET Scan
Number analyzed (Participants) | 173
Number analyzed (Unbiopsied Lesions) | 2057
percentage of lesions | 98

ADVERSE EVENTS:
Time Frame: up to 5 years
Arm/Group | PET Scan
All-Cause Mortality (participants affected / at risk) | 156/173
Serious Adverse Events (participants affected / at risk) | 2/173
Other Adverse Events (participants affected / at risk) | 0/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PET Scan (N=173)
Confusion (Psychiatric disorders) | 1
Fatigue (General disorders) | 1
Renal Failure (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-04-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT00002981/Prot_SAP_000.pdf